CLINICAL TRIAL: NCT02331563
Title: Adjuvant Effect of Dexmedetomidine for the Ultrasound Guided Transversus Abdominis Plane Block in Patients Undergoing Laparascopic Cholecystectomy: a Randomized Controlled Clinical Trial.
Brief Title: Adjuvant Effect of Dexmedetomidine in Ultrasound (USG) Guided Transvers Abdominis Plane Block
Acronym: USG
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: patients should have assurance to attend this study, money is the main problem
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Ferda Yaman, assist prof dr, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20.10.2014/24/07
Record Dates: First submitted 2015-01-01; First posted 2015-01-06 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-01

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: dexmedetomidine
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine; Bupivacaine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5% bupivacaine (Experimental): group 1 receiving TAP block with 0.25% bupivacaine 20 ml for each side of abdomen Bupivacaine is a local anaesthetic agent. transvers abdominis plane block with %0.5 Bustesin which is diluated with normal saline
  Interventions: Drug: 0.25 % bupivacaine
- dexmedetomidine added bupivacaine (Active Comparator): group II receiving TAP block with 0.25% bupivacaine + 0.5 mcg/kg dexmedetomidine each side of abdomen
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — ultrasound guided transvers abdominis plane block
  Other Names: precedex
  Arms: dexmedetomidine added bupivacaine
Drug: 0.25 % bupivacaine — ultrasound guided transvers abdominis plane block
  Other Names: 0.5% Marcaine
  Arms: 0.5% bupivacaine

SUMMARY:
A total of 60 adult patients American Society of Anesthesiologists physical status I,II, III were randomized to Group B (n = 30) receiving TAP block with 0.25% bupivacaine and Group D (n = 30) with 0.5 mcg/kg dexmedetomidine added to 0.25 % bupicavaine followed by general anaesthesia. Total local anaesthetic volume was standardised with 20 ml each sides of the abdomen. Hemodynamic responses to surgical incision and intraoperative fentanyl consumption were noted. Visual analog scale (VAS) scores were assessed on the emergence, at 1, 2, 3, 4, 5, 6 and 24 h. Time to first rescue analgesic (when VAS ≥4 cm or on demand), duration of postoperative analgesia, incidence of postoperative nausea-vomiting were also noted.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block has been shown to provide postoperative pain relief following various abdominal and inguinal surgeries. The aim of this randomised controlled trial was to assess the effect of transversus abdominis plane (TAP) blocks on opioid requirements and median hospitai stay, postoperative nause and vomitting in patients undergoing laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* The patients undergoing laparascopic cholecystectomy

Exclusion Criteria:

* Story of allergy to bupivacaine and dexmedetomidine
* The surgery preceeded to laparatomy
* Recent abdominal operation history

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
opioid requirement | 24 hr
  postoperative relief

SECONDARY OUTCOMES:
postoperative nause and vomiting | 24 hrs
  patient relief

CONTACTS AND LOCATIONS:
Overall Officials: Ferda Yaman, assist prof, Principal Investigator — Kırıkkale University School of Medicine
Locations (1):
- Kırıkkale University School of Medicine Department of Anaesthesiology and Reanimation, Kırıkkale, Yahşihan, Turkey (Türkiye)